CLINICAL TRIAL: NCT05802498
Title: IR3MA Parkinson Cyclone in Life: Innovation, R3 Rehabilitation - Resonance - RTD Fluxgate Sensor, Multidisciplinary Approach
Brief Title: Rehabilitation in Parkinson Disease Cyclone in Life
Acronym: IRMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I.R.M.A.
Record Dates: First submitted 2023-03-15; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2020-07

CONDITIONS: Parkinson Disease; Physical Disability
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control GROUP (No Intervention): This group will perform 8 continuous weeks of treatment, 5 days a week, for a total of 180 minutes, including muscle stretching, joint range increase with passive and active assisted mobilization sessions of the scapulohumeral and pelvic girdles. Motor coordination exercises. Postural exercises with exercises for trunk control in sitting and standing positions with feedback and feed-forward techniques. gait training; gait training; proprioceptive exercises and exercises to maintain static and dynamic balance in monopodalica; strengthening of trunk muscles; postural exercises, muscle relaxation/stretching, release of the tracks; re-education in postural passages and transfers with fall prevention strategies.
- irma group (Experimental): This group will perform 8 continuous weeks of treatment, 5 days a week, for a total of 180 minutes, including muscle stretching, increasing joint range with assisted passive and active mobilisation sessions of the scapulohumeral and pelvic girdles. Motor coordination exercises. Postural exercises with exercises for trunk control in sitting and standing with feedback and feed-forward technique. Gait training; gait training; proprioceptive exercises and static and dynamic balance maintenance in monopodalics; trunk muscle strengthening; postural exercises, muscle relaxation/relaxation, caterpillar release; re-education in postural transitions and transfers with fall prevention strategies. Prior to neuromotor rehabilitation treatment, the subjects will undergo rehabilitation training using the NIRVANA augmentative reality system.
  Interventions: Device: IRMA

INTERVENTIONS:
Device: IRMA — For patients in an advanced state of illness, advanced neuromotor rehabilitation treatment included 1) robot therapies, 2) specific water courses (e.g. walking pools, hydrokinesiotherapy pools, etc.), 3) advanced cognitive treatments (e.g. virtual reality courses); 4) augmentative immersive therapy in a virtual environment; 5) courses also dedicated to social reintegration and inclusive activities (theatre-therapy, art-therapy, dance-therapy, agro-therapy, etc.).
  Arms: irma group

SUMMARY:
Comparison of two rehabilitation protocols in patients with Parkinson's disease and, therefore, identification of innovative rehabilitation protocols of proven and validated efficacy, through which it is possible to achieve:

* Improved joint function and gait pattern
* Reduction of the risk of falling or reduction of energy expenditure during physiological gait

Evaluation of the increase in maximal effort tolerance

· Improved cognitive performances

Evaluation of the impact on the quality of life of the patient and family members

Identification of morpho-functional markers predictive of clinical and rehabilitative out-come through neuroimaging study.

DETAILED DESCRIPTION:
rehabilitation protocols in patients with Parkinson's disease and, therefore, identification of innovative rehabilitation protocols of proven and validated efficacy, through which it is possible to achieve:

Improved joint function and gait pattern Reduction of the risk of falling or reduction of energy expenditure during physiological gait Evaluation of the increase in maximal effort tolerance

· Improved cognitive performances

Evaluation of the impact on the quality of life of the patient and family members

Identification of morpho-functional markers predictive of clinical and rehabilitative out-come through neuroimaging study.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn & Yahr between 2.0 and 3.0;
* No need for a walking aid;
* Mini-Mental State Examination (MMSE) score >24;
* Effective dopaminergic pharmacological control;
* Absence of other relevant neurological comorbidities;
* Absence of postural deformities (and/or Pisa syndrome);
* Absence of severe cardiological pathologies (exertional angina, severe decompensation).
* Ability to travel to the rehabilitation treatment site independently or with support

Exclusion Criteria:

* presence of Deep Brain Stimulation (DBS);
* presence of severe heart and/or lung disease;
* presence of therapeutic regimen in the definition phase;
* impaired joint and/or motor function to follow a proposed rehabilitation treatment programme
* contraindications to performing MRI scans
* undergoing rehabilitation therapy in the 3 months preceding enrolment.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | 8 weeks
  The Berg Balance Scale is a scale for assessing balance and the risk of falling

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro Neurolesi "Bonino-Pulejo", Messina, Italy

IPD SHARING:
Plan to Share IPD: No
corresponding author